CLINICAL TRIAL: NCT07081997
Title: A Phase 3, Multicenter, Single Arm, Open-Label Trial Investigating the Safety, Tolerability and Efficacy of Palopegteriparatide Administered Subcutaneously Daily at Doses Greater Than 30 µg/Day in Adult Participants With Hypoparathyroidism
Brief Title: A Phase 3 Clinical Trial to Investigate the Safety and Efficacy of Palopegteriparatide at Doses Greater Than 30 μg/Day in Adult Participants With Hypoparathyroidism
Acronym: PaTHway60
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ascendis Pharma Bone Diseases A/S (Industry)
Responsible Party: Sponsor
Organization: Ascendis Pharma A/S (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASND0052
Record Dates: First submitted 2025-07-22; First posted 2025-07-24 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Hypoparathyroidism; Endocrine System Diseases; Parathyroid Diseases
Keywords: Hypoparathyroidism; Parathyroid Hormone; TransCon PTH; PTH(1-34); Prodrug; Sustained Release; Parathyroid Hormone Replacement Therapy; Palopegteriparatide
MeSH Terms: conditions — Hypoparathyroidism; Endocrine System Diseases; Parathyroid Diseases

STUDY DESIGN:
Intervention Model Description: Open label single-arm multi-center
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Palopegteriparatide (Experimental): Palopegteriparatide at doses at or greater than 30 mcg delivered once daily by subcutaneous injection and titrated to an optimal dose
  Interventions: Combination Product: Palopegteriparatide

INTERVENTIONS:
Combination Product: Palopegteriparatide — Palopegteriparatide is supplied as a solution with a concentration of 0.3 mg/mL in a single-patient-use prefilled pen intended for subcutaneous injection.
  Other Names: Yorvipath

SUMMARY:
This trial has a duration of 78 weeks and will include adult participants already on treatment with palopegteriparatide at doses at or greater than 30 mcg/day. All participants will receive subcutaneous palopegteriparatide during the trial and will be individually and progressively titrated to an optimal dose at pre-specified dose levels. The primary purpose of the trial is to provide additional evidence of treatment effect and safety of palopegteriparatide at doses greater than 30 mcg/day in adults with hypoparathyroidism. The trial will be conducted in the US.

ELIGIBILITY:
Inclusion criteria:

1. Males and females, ≥18 years of age at the time of providing informed consent
2. Participants with postsurgical chronic hypoparathyroidism (HP), or auto-immune, genetic, or idiopathic HP, for at least 26 weeks
3. Receiving doses of palopegteriparatide at or above 30 µg/day

   For individuals receiving 30 µg/day: evidence that dose is insufficient to keep serum calcium in the normal range, defined as:

   Documented hypocalcemia within 12 weeks prior to Screening; and/or Standing dose of calcitriol ≥0.25 μg/day, and / or (elemental) calcium ≥1500 mg/day (e.g., calcium citrate, calcium carbonate etc.) for at least 4 weeks prior to Screening

   For individuals receiving 33 µg/day or greater: no requirement for documented hypocalcemia or minimum doses of calcitriol or elemental calcium
4. Confirmation of laboratory parameters (Central and Local) within 2 weeks of screening visit:

25(OH) vitamin D levels of 20 - 80 ng/mL (49 - 200 nmol/L) and Magnesium level in the normal range, or just below the normal range i.e.: ≥1.3 mg/dL (≥0.53 mmol/L) and Albumin-adjusted or ionized sCa level in the normal range or just below the normal range

* Albumin-adjusted sCa 7.8 - 10.6 mg/dL (or 1.95 - 2.64 mmol/L)
* Ionized sCa 4.40 - 5.29 mg/dL (1.10 - 1.32 mmol/L)

  5. BMI 17- 40 kg/m2 at Screening

  6. If ≤25 years of age, radiological evidence of epiphyseal closure based on locally interpreted X-ray of non-dominant wrist and hand

  7. eGFR ≥30 mL/min/1.73 m2 during Screening using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula

Exclusion criteria

1. Impaired responsiveness to PTH (pseudohypoparathyroidism), which is characterized as PTH-resistance, with elevated PTH levels in the setting of hypocalcemia
2. Any disease that might affect calcium metabolism or calcium-phosphate homeostasis or PTH levels other than HP
3. Use of loop diuretics, phosphate binders (other than calcium supplements), digoxin, lithium, methotrexate, biotin >30 µg/day, or systemic corticosteroids (other than as replacement therapy)
4. Use of thiazide diuretic within 4 weeks prior to the 24-hour urine collection scheduled to occur within 1 week prior to Visit 1
5. Use of PTH-like drugs other than palopegteriparatide (whether commercially available or through participation in an investigational trial), including PTH(1-34), or other N-terminal fragments, analogs of PTH or PTH-related protein, or PTH1R biased agonists within 4 weeks prior to Screening
6. Use of drugs known to influence calcium and bone metabolism within 12 weeks prior to Screening
7. Use of osteoporosis therapies other than bisphosponate known to influence calcium and bone metabolism within 2 years prior to Screening. Note: use of bisphosphonate (oral or intravenous [IV] is not exclusionary
8. Non-hypocalcemic seizure disorder with occurrence of a seizure within 26 weeks prior to Screening.
9. Increased risk for osteosarcoma
10. Women who are pregnant, intend to become pregnant, or are lactating
11. Male who has a female partner who intends to become pregnant or is of childbearing potential and is unwilling to use adequate contraceptive methods during the trial
12. Diagnosed drug or alcohol dependence within 3 years prior to Screening
13. Chronic or severe cardiac disease within 26 weeks prior to Screening
14. Cerebrovascular accident within 5 years prior to Screening.
15. Within 26 weeks prior to Screening: acute colic due to nephrolithiasis, or acute gout
16. Participation in any other interventional trial in which receipt of investigational drug or device other than palopegteriparatide occurred within 8 weeks (or within 5.5 times the half-life of the investigational drug) (whichever comes first) prior to Screening.
17. Known allergy or sensitivity to PTH or any of the excipients [metacresol, mannitol, succinic acid, NaOH/(HCl)] of the investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy - Primary endpoint | 26 weeks
  The proportion of participants with:
  Albumin-adjusted serum calcium (sCa) measured within 4 weeks prior to and on the Week 26 visit within the normal range (8.3-10.6 mg/dL); and independence from active vitamin D; and independence from therapeutic doses of calcium; and no increase in prescribed investigational product within 4 weeks prior to Week 26 visit.

CONTACTS AND LOCATIONS:
Overall Officials: Claus Strange, Study Director — Ascendis Pharma A/S

IPD SHARING:
Plan to Share IPD: No